CLINICAL TRIAL: NCT04454151
Title: Azithromycin Treatment for Readthrough of APC Gene Stop Codon Mutations in Familial Adenomatous Polyposis
Acronym: FAP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, michal roll, director, R&D Division, Tel-Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-19-RK-682-CTIL
Record Dates: First submitted 2020-02-04; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Familial Adenomatous Polyposis
Keywords: Azithromycin Familial Adenomatous Polyposis (FAP) APC gene nonsense mutations
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Azithromycin (Experimental): 1x250
  Interventions: Drug: Azithromycin Tablets

INTERVENTIONS:
Drug: Azithromycin Tablets — given PO Azithromycin 250 mg X1 daily, for 4 months, followed by a non-treatment follow-up period of 12 month.

SUMMARY:
Colorectal cancer (CRC) is a leading cause for cancer related mortality in the western world with a lifetime risk of 6%. Etiology is complex, while genetic background significantly affects the risk. Around one third of all genetic disorders as well as most cases of Familial Adenomatous Polyposis (FAP) and a large proportion of all sporadic CRC cases occur as a result of premature nonsense mutations (creating a stop codon) in an individual's adenomatous polyposis coli (APC) gene. Nonsense mutations are single-point alterations in the DNA that prematurely halt the protein translation process, producing a shortened, nonfunctional protein. In many of these cases, if the cell can be 'persuaded' to ignore the premature stop codon signal, the resulting protein may be able to ameliorate or stop the disease.

Recently, members of the aminoglycoside family of antibiotics have been found to induce ribosomal read-through of nonsense mutations, leading to expression of a full length, functional protein. Investigators have recently shown that members of the aminoglycoside and macrolide antibiotic families can induce read-through of the nonsense mutations in the APC gene and lead to reduced oncogenic phenotypes in CRC cells and in different mice models.

The aim of this project is to determine the ability of the macrolide antibiotic-Azithromycin to induce read-through of the nonsense mutations in the APC gene and to induce expression of a full length, functional APC protein in patients suffering from FAP and to tests its effect on adenoma number and size and on desmoid tumors in these patients. The future goal is to maximize the effect of stop-codon suppressors on APC while minimizing side effects.

In this study the investigators will select FAP patients which carry APC nonsense mutations, treat them with Azithromycin PO for 4-6 months and examine colonic and duodenal adenomas as well as abdominal desmoid tumors, that will be documented before during and after treatment. In parallel, investigators will test polyp, adenoma and desmoid tissue samples as well as blood samples from these patients for changes in expression levels of the APC protein and related oncogenic markers.

Suppression of nonsense mutations within the APC gene should be of benefit for patients suffering from FAP, attenuated FAP or multiple adenomas and for patients with advanced or diffuse CRC. Furthermore, given the rapid progress being made in the identification of different nonsense mutations in human genes that lead to mostly non-curable disease, the identification of clinically approved compounds that suppress nonsense mutations and that can be administered long-term without significant side effects would open new venues in the treatment of genetic human diseases that arise from pre-mature stop codons in important coding sequences.

Immediate goal: establish the ability of Azithromycin to read-through APC nonsense mutation in FAP patients. The read-through effect of Azithromycin will be clinically tested by counting and measuring the number and size of both colonic and duodenal adenomas before and over treatment and by measuring the size of known desmoid tumors. Samples of the adenomas and desmoid tumors will be tested by western blot, immunofluorescence and immunohistochemistry for restoration of APC expression and changes in oncogenic markers. These experiments should be conducted within 6 month.

Long term objective:

1. Determine the lowest dose of Azithromycin that can inhibit growth of colonic neoplasia and CRC in patients expressing a truncated APC protein due to nonsense mutations.
2. Examine the ability of a panel of additional macrolide antibiotics to induce APC nonsense mutation suppression using in-vitro methods. Investigators will focus on macrolide antibiotics that are currently in clinical use and are administrated for long terms. These objectives should take around 4 month and will be conducted in parallel.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18Y who carry a hereditary APC nonsense mutation as identified by APC sequencing. The sequencing is performed by the Israeli Health Ministry's certified genetic lab and the mutation is approved by a certified geneticist or genetic counsel as a nonsense stop codon mutation.
2. Presence of at least 3 polyps, among which at least 1 is equal or larger than 3 mm. Polyp location is in the intact colon, in the rectal remnant in patients that underwent subtotal colectomy with ileorectal anastomosis or in the ileoanal pouch in patients who underwent total proctocolectomy with ileoanal pouch anastomosis.
3. Reading and signing the informed consent form.

Exclusion Criteria:

1. Age < 18Y
2. Pregnancy or planning pregnancy in the near future
3. Hypersensitivity to the active substance, erythromycin, any macrolide, ketolide antibiotic, soya lecithin and/or any of the following Microcrystalline cellulose, Pregelatinised maize starch, Sodium starch glycolate Type A, Colloidal anhydrous silica, Sodium laurilsulfate, Magnesium stearate, Polyvinyl alcohol, Titanium dioxide (E 171), Talc, Soya Lecithin, Xanthan Gum.
4. Chromic Hypokalemia or hypomagnesemia
5. Significant personal or family history of ventricular arrhythmia
6. Long QT interval per ECG, or consumption of drugs that may cause prolonged QT.
7. Molecular evidence of variant for the congenital long QT syndrome
8. Advanced polyp or desmoids tumor that requires immediate treatment.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of changes in number of adenomas measured by upper endoscopy | After 8,16 weeks and 12 months
  Change in number of adenomas from baseline will be measured by endoscopic and histological evaluation. response will be tested by upper and lower endoscopies after 8 ,16-20 weeks and 12 months of treatment
Evaluation of changes in size of adenomas measured by upper endoscopy | After 8,16 weeks and 12 months
  Change in size of adenomas from baseline will be measured by endoscopic and histological evaluation. response will be tested by upper and lower endoscopies after 8 ,16-20 weeks and 12 months of treatment

SECONDARY OUTCOMES:
Evaluation of changes in number of adenomas measured by lower endoscopy | After 8,16 weeks and 12 months
  Change in number of adenomas from baseline will be measured by endoscopic and histological evaluation. response will be tested by upper and lower endoscopies after 8 ,16-20 weeks and 12 months of treatment.
Evaluation of changes in size of adenomas measured by lower endoscopy | After 8,16 weeks and 12 months
  Change in size of adenomas from baseline will be measured by endoscopic and histological evaluation. response will be tested by upper and lower endoscopies after 8 ,16-20 weeks and 12 months of treatment.

OTHER OUTCOMES:
Evaluation of changes in number of desmoid tumors | At the begining of the trial (before treatment) and at the end of the treatment (after 4-6 months)
  Desmoids imaging (US or CT or MRI) will be performed to determine the number at the begining of the study and to evaluate the change from baseline after 4-6 months of treatment.
Evaluation of changes in size of desmoid tumors | At the begining of the trial (before treatment) and at the end of the treatment (after 4-6 months)
  Desmoids imaging (US or CT or MRI) will be performed to determine the size at the begining of the study and to evaluate the change from baseline after 4-6 months of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Sourasky medical center (Ichilov), Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided